CLINICAL TRIAL: NCT05255393
Title: RELEVANT Prevalence of Patient-Reported Lymphedema Following Surgical Management of Cervical or Vulvar Cancer
Brief Title: Survey on Lymphedema After Sentinel Lymph Node Biopsy in People With Cervical or Vulvar Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-002
Record Dates: First submitted 2022-02-16; First posted 2022-02-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer; Vulvar Cancer
Keywords: Questionnaire; Sentinel Lymph Node Biopsy; Lymphedema; 22-002
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Lymphedema | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard lymphadenectomy(LND) with sentinel lymph node mapping (SLN): Patients will receive up to two mailings or messages and two phone calls if they do not respond. Self-addressed, stamped envelopes will be provided for return of questionnaires.
  No other interventions are planned.
  Interventions: Other: Questionnaires
- Standard lymphadenectomy(LND) alone: Patients will receive up to two mailings or messages and two phone calls if they do not respond. Self-addressed, stamped envelopes will be provided for return of questionnaires.
  No other interventions are planned.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — A 13-item questionnaire specific to LEL, developed and validated by investigators at the Mayo Clinic.
  The EORTC QLQ-C30 is a 30-item questionnaire designed to assess the quality of life of cancer patients.
  The EORTC Quality of Life - Cervical Cancer Module.

SUMMARY:
The purpose of this study is to collect information that may identify people who are at risk of developing lower extremity lymphedema (LEL) after sentinel lymph node biopsy (SLN) during surgery for early-stage vulvar or cervical cancer, and to improve the quality and accuracy of the information that is given to people who have this procedure.

Please note that, during this study, the researchers will collect information from a questionnaire completed by people who had SLN and LND+/- SLN during surgery for early-stage cervical or vulvar cancer. No form of treatment will be provided as part of the study, and no investigational tests or procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Presented to MSK with newly diagnosed early-stage cervical cancer of any histologic profile or early stage vulvar cancer of any histologic profile.

  °Early stage: Stage 1-2
* Underwent primary surgery at our institution between January 2006 and January 2022.
* Alive at the time of study activation
* English comprehension
* Capable of providing informed consent

Exclusion Criteria:

* Had documented macroscopic evidence of metastatic disease at the time of initial diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cervical or Vulvar Cancer
Study Population: All patients in the GYN DMT's cervical cancer and vulvar cancer databases
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
prevalence of patient-reported lower extremity lymphedema | 1 year
  Prevalence will be measured using the 13-item questionnaire as reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Leitao, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm